CLINICAL TRIAL: NCT04109235
Title: IS SHORT-DURATION, HIGH-INTENSITY-INTERVAL TRAINING (HIIT) SUPERIOR TO POPULATION-BASED MODERATE-INTENSITY PHYSICAL ACTIVITY GUIDELINES FOR INDIVIDUALS WITH TYPE 2 DIABETES? A PILOT STUDY
Brief Title: Family Health Team High-Intensity Interval Training
Acronym: FHT HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: East Elgin Family Health Team (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111930
Record Dates: First submitted 2019-09-12; First posted 2019-09-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes
Keywords: HbA1C; virtual care; blood glucose; physical activity; HIIT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Masking Description: One of the investigators, Justine Horne, will be blinded to group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population-Based Physical Activity (PA) Advice (Active Comparator): This PA intervention will be primarily self-directed by the patients themselves. Each participant will receive a 1-page double-sided handout detailing their PA protocol. Participants in this arm will receive a CSEP handout (page 4&5 from: http://csep.ca/CMFiles/Guidelines/CSEP_PAGuidelines_0-65plus_en.pdf) detailing their PA recommendations.Participants will be instructed to follow their PA protocol, while noting down which days they completed the PA using a log booklet provided to them by Dr. Fernando (their family physician). Participants will be provided with the phone number for a research assistant who is a lifestyle coach and co-investigator on this trial. If participants have questions about their PA protocol, the research assistant will respond to these over the phone.
  Interventions: Other: Population-Based Physical Activity (PA) Advice
- High-Intensity Interval Training Physical Activity (PA) Advice (Experimental): This PA intervention will be primarily self-directed by the patients themselves. Each participant will receive a 1-page double-sided handout detailing their PA protocol. Participants in this arm will receive a High-Intensity-Interval-Training (HIIT) handout (developed based on research from Dr. Martin Gibala) detailing their PA recommendations. Participants will be instructed to follow their PA protocol, while noting down which days they completed the PA using a log booklet provided to them by Dr. Fernando (their family physician). Participants will be provided with the phone number for a research assistant who is a lifestyle coach and co-investigator on this trial. If participants have questions about their PA protocol, the research assistant will respond to these over the phone.
  Interventions: Other: High-Intensity Interval Training Physical Activity (PA) Advice

INTERVENTIONS:
Other: High-Intensity Interval Training Physical Activity (PA) Advice — This PA intervention will be primarily self-directed by the patients themselves. Each participant will receive a 1-page double-sided handout detailing their PA protocol. Participants in this arm will receive a High-Intensity-Interval-Training (HIIT) handout (developed based on research from Dr. Martin Gibala) detailing their PA recommendations. Participants will be instructed to follow their PA protocol, while noting down which days they completed the PA using a log booklet provided to them by Dr. Fernando (their family physician). Participants will be provided with the phone number for a research assistant who is a lifestyle coach and co-investigator on this trial. If participants have questions about their PA protocol, the research assistant will respond to these over the phone.
  Arms: High-Intensity Interval Training Physical Activity (PA) Advice
Other: Population-Based Physical Activity (PA) Advice — This PA intervention will be primarily self-directed by the patients themselves. Each participant will receive a 1-page double-sided handout detailing their PA protocol. Participants in this arm will receive a CSEP handout (page 4&5 from: http://csep.ca/CMFiles/Guidelines/CSEP_PAGuidelines_0-65plus_en.pdf) detailing their PA recommendations.Participants will be instructed to follow their PA protocol, while noting down which days they completed the PA using a log booklet provided to them by Dr. Fernando (their family physician). Participants will be provided with the phone number for a research assistant who is a lifestyle coach and co-investigator on this trial. If participants have questions about their PA protocol, the research assistant will respond to these over the phone.
  Arms: Population-Based Physical Activity (PA) Advice

SUMMARY:
With the rapid shift to virtual care, this pilot study aims to determine the feasibility of prescribing low-duration, interval-based training through virtual care. If successful, this study will inform a larger randomized control trial to determine if the prescription of low-duration interval-based training improves chronic disease through the measurement of hemoglobin A1C (HbA1C), and weight to a greater extent than the general guideline to aim for 150 minutes of PA weekly.

DETAILED DESCRIPTION:
Dr. Fernando will invite patients to participate in this trial during their virtual diabetes appointments at the East Elgin Family Health Team (EEFHT). Participants will be randomized 1:1 using computer-generated randomization software to receive either a population-based, standard activity intervention (control group) or a high-intensity interval training (HIIT) intervention, which they will complete on their own time, at the location of their choosing (at home, gym, outside, or elsewhere). Data will be collected at baseline (T1), and participants will be followed up after 3 months (T2) and 6 months (T3). All data acquisition is from standard of care (i.e. patients are already seen every 3 months for diabetes visits). Data collection at T1, T2 and T3 will include:

* Weight and Height (measured using the Health-O-Meter weigh scale, used to calculate BMI)
* Minutes of PA (self-reported by participants using the log books designed for this study)
* HbA1C (requisition will be provided by Dr. Fernando. Patients will be exempt from completing the baseline HbA1C if they have had a HbA1C measurement in the past 30 days & the patient has not made significant lifestyle changes or had any blood glucose medications changed; in this case, the measurement completed in the past 30 days will be used as the baseline measure)
* Blood glucose and blood pressure medications

ELIGIBILITY:
Inclusion Criteria:

* adults, at least 18 years of age
* non-pregnant
* having a diagnosis of type 2 diabetes in accordance with the 2018 Diabetes Canada Clinical Practice Guidelines
* capable of consenting
* deemed capable and safe to exercise by their physician (Dr. Fernando)
* without a medical history of myocardial infarction in the past three months.

Exclusion Criteria:

* < 18 years of age
* pregnant
* not having a type 2 diabetes diagnosis
* having a medical history of myocardial infarction in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C | 3-month and 6-month follow-up
  Glycosylated Hemoglobin measured at lab

SECONDARY OUTCOMES:
Weight | 3-month and 6-month follow-up
  self-reported by participants using home scale
Physical Activity (minutes per week) | 3-month and 6-month follow-up
  self-reported by participants using the log books designed for this study

CONTACTS AND LOCATIONS:
Locations (1):
- East Elgin Family Health Team, Aylmer, Ontario, Canada